CLINICAL TRIAL: NCT02089425
Title: An Efficacy and Safety Study for the Treatment of Mild to Moderate Acute Pain Associated With Ankle Strain or Sprain.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim futility analysis
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-103-IP-3.01US
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Acute Pain From Ankle Sprain or Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo patch: 0% indomethacin
  Interventions: Drug: Placebo
- K-103-IP (Experimental): K-103-IP: 0.5% indomethacin
  Interventions: Drug: K-103-IP

INTERVENTIONS:
Drug: K-103-IP
  Arms: K-103-IP
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled, parallel group study to assess the efficacy and safety of K-103-IP compared with placebo patch for treatment of mild to moderate acute pain associated with ankle strain or sprain.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide informed consent before any study specific evaluation is performed.
* Subject is male or female aged 18 to 70 years, inclusive.
* Subject has a grade 1 (mild functional impairment) or grade 2 (moderate functional impairment) ankle strain or sprain that occurred within 48 hours before the Screening visit.
* Subject has pain intensity upon monopodal weight bearing of 5 to 8, inclusive, measured by an 11 point nominal rating scale (NRS), plus pain intensity score at rest that is less than upon monopodal weight bearing.

Exclusion Criteria:

* Subject has a grade 3 (severe functional impairment) strain or sprain, bilateral strain or sprain, or concomitant fracture or wound at the site of the strain or sprain.
* Subject has had an ankle strain or sprain to the same foot within 6 months before the Screening visit.
* Subject has received topical analgesic medication within 24 hours before the Screening visit.
* Subject has applied ice or compression to the injured area within 2 hours before the Screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference(SPID) 0-72 | 72 Hours

SECONDARY OUTCOMES:
Mean change from Baseline in pain intensity difference (PID) | 168 Hours

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Anaheim, California
  - El Cajon, California
  - Encinitas, California
  - Los Angeles, California
  - Ventura, California
  - Boynton Beach, Florida
  - Daytona Beach, Florida
  - Doral, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Oldsmar, Florida
  - Orlando, Florida
  - Port Orange, Florida
  - Chicago, Illinois
  - Overland Park, Kansas
  - Owensboro, Kentucky
  - Towson, Maryland
  - Rochester, Michigan
  - St Louis, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Atco, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Mooresville, North Carolina
  - Morganton, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Willoughby, Ohio
  - Gresham, Oregon
  - Rapid City, South Dakota
  - Jackson, Tennessee
  - Memphis, Tennessee
  - Smyrna, Tennessee
  - Austin, Texas
  - Boerne, Texas
  - El Paso, Texas
  - Houston, Texas
  - Bountiful, Utah
  - Salt Lake City, Utah